CLINICAL TRIAL: NCT05770700
Title: Effectiveness and Safety of Implantable Neurostimulation Systems for the Treatment of Chronic Refractory Pain in Spain: Prospective Multicenter Study From the Spanish Pain Society Registry (STIM-RENASED)
Brief Title: Effectiveness and Safety of Implantable Neurostimulation Systems for Chronic Pain: A Spanish Multicenter Study (STIM-RENASED)
Acronym: STIM-RENASED
Status: Recruiting | Type: Observational
Sponsor: Sociedad Espanola del Dolor (Other)
Responsible Party: Sponsor
Other Study IDs: PI 238/22
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain
Keywords: Spinal cord stimulation; Dorsal root ganglion stimulation; Peripheral nerve stimulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic pain is a prevalent condition that negatively affects patients' quality of life. Implantable neurostimulation therapies have been proposed as a treatment option for chronic pain. However, real-world data on the effectiveness and safety of these therapies in Spain are scarce. This study aims to obtain real-world data on the effectiveness and safety of implantable stimulation systems for chronic pain treatment in Spain.

DETAILED DESCRIPTION:
All Spanish hospitals that implant neurostimulation systems for pain treatment will be invited to participate in the study. Patients will be recruited before the procedure, and before providing data to the registry, the study will be explained to them, and they will sign an informed consent form. Demographic data related to the pathology and procedure will be collected. Follow-up will be conducted at six and twelve months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Chronic refractory pain patients candidates for treatment with an implantable neurostimulation system.
* Accept to participate in the study and sign informed consent.

Exclusion Criteria:

* Patients in whom it would be difficult to complete follow-up.
* Insufficient understanding of the Spanish language.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic refractory pain who are candidates for treatment with a implantable neurostimulation system.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with at least 50 % pain relief in the area of their predominant pain at one year. | Twelve months
  Percentage of patients who experience a reduction of at least 50% in the intensity of their predominant pain compared to the initial value, assessed twelve months after the implantation of the neurostimulation system. Pain intensity will be measured using an 11-point Numeric Pain Rating Scale (NPRS), with a range from 0 (no pain) to 10 (maximum pain possible)

SECONDARY OUTCOMES:
Percentage of patients with at least 50 % pain relief in the area of their predominant pain at six months. | Six months
  Percentage of patients who experience a reduction of at least 50% in the intensity of their predominant pain compared to the initial value, assessed six months after the implantation of the neurostimulation system. Pain intensity will be measured using an 11-point Numeric Pain Rating Scale (NPRS), with a range from 0 (no pain) to 10 (maximum pain possible)
Percentage of patients with at least 50 % pain relief in the area of their non-predominant pain at one year. | Six and twelve months
  Percentage of patients who experience a reduction of at least 50% in the intensity of their non-predominant pain compared to the initial value, assessed six and twelve months after the implantation of the neurostimulation system. Pain intensity will be measured using an 11-point Numeric Pain Rating Scale (NPRS), with a range from 0 (no pain) to 10 (maximum pain possible)
Compared change from baseline on health-related quality of life scores (EQ Index) | Six and twelve months
  The impact of the treatment on the patient's health-related quality of life will be evaluated using the EQ-5D-5L questionnaire at six and twelve months after implantation. The EQ-5D-5L assesses quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is scored on a scale of 1 (no problems) to 5 (extreme problems), generating a 5-digit code that corresponds to the patient's health status.
Patient Global Impression of Improvement | Six and twelve months
  Assessment of clinical global impression of improvement using the PGI-I scale at six and twelve months after implantation of the neurostimulation system. The PGI-I score ranges from 1 (Very much better) through to 7 (Very much worse). The lower the score, the better the improvement.
Patient Satisfaction | Six and twelve months
  Percentage of implanted subjects satisfied with the treatment at six and twelve months after the implantation of the neurostimulation system. defined as indicating: "since the start of the therapy has the pain improved? yes/no", "Are you satisfied with the treatment?" yes/no or "would you agree to the treatment again?" yes/no
Number of Adverse Events as a Measure of Safety | Six and twelve months
  Number and percentage of patients with adverse effects related to therapy at six and twelve months after implantation of the neurostimulation system.

CONTACTS AND LOCATIONS:
Locations (16):
- Spain (16):
  - Hospital FREMAP Majadahonda, Majadahonda, Madrid
  - Complejo Hospitalario Universitario de Cartagena, Cartagena, Murcia
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Regional Univeristario de Málaga, Málaga
  - Complexo Hospitalario Univeritario de Ourense, Ourense
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo